CLINICAL TRIAL: NCT01373580
Title: A Prospective, Multinational Multicenter Clinical Trial to Evaluate the Safety and Effectiveness of the ReVision Optics, Inc. PresbyLens Corneal Inlay for the Improvement of Near Vision in Presbyopic Subjects With MRSE From -0.50 to +1.00
Brief Title: A Clinical Trial to Evaluate a Corneal Inlay for the Improvement of Near Vision in Presbyopic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReVision Optics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P09-0003
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Presbyopia
Keywords: presbyopia; LASIK; loss of accommodation; Emmetrope
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raindrop (Experimental): A single-arm study to evaluate the effectiveness of a 2 mm corneal inlay (Raindrop Near Vision Inlay) for the treatment of presbyopia (age-related near vision loss). The anterior curvature of the cornea is re-shaped after implanting the Raindrop Near Vision Inlay in the non-dominant eye under a femtosecond laser flap to improve near vision.
  Interventions: Device: The Raindrop Near Vision Inlay

INTERVENTIONS:
Device: The Raindrop Near Vision Inlay — The Raindrop Near Vision Inlay is implanted in the cornea for treatment of presbyopia
  Other Names: Presbylens

SUMMARY:
This study will be a prospective, multicenter clinical trial in which a total of 400 subjects will be enrolled. All subjects will be followed over a 36 month time frame with a maximum of 15 clinical sites participating. Qualified subjects will provide informed consent for entry into the study.

DETAILED DESCRIPTION:
The loss of near vision and the ability to perform tasks that require near vision is part of the normal aging process. This natural transformation in the eye occurs as a result of the loss of accommodation of the crystalline lens, a condition known as presbyopia. Presbyopia, characterized by a progressive, age-related loss of accommodation (i.e., the lens ability to focus clearly over a wide range of distances), is most prevalent of all visual deficiencies, affecting 100% of the population over the course of a normal life span. Loss of accommodation begins early in life and, for an emmetropic eye, generally culminates in a complete loss of functional near vision.

ReVision Optics has developed the Raindrop corneal inlay for the correction of near vision. The Raindrop is a 2mm corneal inlay, as small as a pinhead, thinner than a human hair and about 1/500th of a droplet of water. The inlay is the same refractive index as the human cornea. The inlay is placed in the non-dominant eye,centered over the pupil after a corneal flap (LASIK)has been made. The Raindrop is expected to provide presbyopic subjects with improvement of near and intermediate vision.

ELIGIBILITY:
Inclusion Criteria:

must be presbyopic adults, needing from +1.50 to +2.50 or reading add must have uncorrected near visual acuity worse than 20/40 and better than 20/200in the eye to be implanted must have an uncorrected distance visual acuity of 20/25 or better in both eyes must have a distance visual acuity correctable to 20/20 in both eyes must have a near visual acuity correctable to 20/20 in both eyes must have a manifest refraction spherical equivalent between -0.50 and +1.00D in the eye to be implanted with no more than 0.75D of refractive cylinder must report stable vision, i.e. no change in distance vision and or MRSE within 0.50D over prior 12 months must discontinue hard or rigid gas permeable lenses for at least 3 weeks and discontinue soft lenses for at least 1 week prior to baseline examination must have a minimum central corneal thickness of >500 microns in the eye to be implanted must have a mesopic pupil < 7.0mm and photopic pupil >3.0mm in the eye to be implanted subjects aged 45 years or younger must have an endothelial cell count

Exclusion Criteria:

Subjects with a difference of >0.75 between the manifest refraction spherical equivalent and the cycloplegic refraction spherical equivalent Subjects with anterior segment pathology, including clinically significant cataracts, in the non-dominant eye Subjects with residual, recurrent, active ocular or uncontrolled eyelid disease, or any corneal abnormality (including endothelial dystrophy, guttata, recurrent corneal erosion, etc.) in the non-dominant eye Subjects with ophthalmoscopic signs of keratoconus (or keratoconus suspect) in the non-dominant eye Subjects with clinically significant dry eyes, as determined by either the presence of greater than mild symptoms of dryness or discomfort or SPK greater than grade 1 Subjects with distorted or unclear mires on topography maps of the non-dominant eye Subjects with macular degeneration, retinal detachment, or any other fundus pathology that would prevent an acceptable visual outcome in the non-dominant eye Subjects who have undergone LASIK surgery in the non-dominant eye Subjects with a history of herpes zoster or herpes simplex keratitis Subjects who have a history of steroid responsive rise in intraocular pressure, pre-operative IOP>21 mm Hg, glaucoma or are a glaucoma suspect Subjects with a history of diagnosed diabetes, autoimmune disease, connective tissue disease, or clinically significant atopic syndrome Subjects on chronic systemic corticosteroids or other immunosuppressive therapy that may affect wound healing, and any immunocompromised subjects Subjects who are using ophthalmic mediation(s) other than artificial tears for treatment of any ocular pathology Subjects using systemic medications with significant ocular side effects Subjects who are pregnant, lactating, or planning to become pregnant during the course of the study Subjects what are participating in any other ophthalmic drug or device studies during the time of this clinical investigation Subjects with known sensitivity to planned study concomitant medications

-

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2010-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven G Slade, M.D., Principal Investigator; Jon G Dishler, MD, Principal Investigator; John Olkowski, M.D., Principal Investigator; Dan B Tran, M.D., Principal Investigator; Ralph Y Chu, M.D., Principal Investigator; Jeffrey Whitman, M.D., Principal Investigator; Robert P Lehmann, M.D., Principal Investigator; Gregory Parkhurst, M.D, Principal Investigator — Unaffilliated; Harvey L Carter, III, M.D., Principal Investigator — Unaffilliated; Paul Dougherty, M.D., Principal Investigator — Unaffilliated; John Hovanesian, M.D., Principal Investigator — Unaffilliated
Locations (11):
- United States (11):
  - Dougherty Laser Vision, Camarillo, California
  - Harvard Eye Associates, Laguna Hills, California
  - Coastal Vision, Newport Beach, California
  - Jon G. Dishler, M.D., Greenwood Village, Colorado
  - Eyesight Hawaai, Honolulu, Hawaii
  - Chu Vision, Bloomington, Minnesota
  - Key-Whitman Eye Center, Dallas, Texas
  - Carter Eye Center, Dallas, Texas
  - Slade and Baker Vision Center, Houston, Texas
  - Lehmann Eye Center, Nacogdoches, Texas
  - NuVision., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitman J, Dougherty PJ, Parkhurst GD, Olkowski J, Slade SG, Hovanesian J, Chu R, Dishler J, Tran DB, Lehmann R, Carter H, Steinert RF, Koch DD. Treatment of Presbyopia in Emmetropes Using a Shape-Changing Corneal Inlay: One-Year Clinical Outcomes. Ophthalmology. 2016 Mar;123(3):466-75. doi: 10.1016/j.ophtha.2015.11.011. Epub 2016 Jan 27. PMID 26804761

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Raindrop
Started | 373
Completed | 317
Not Completed | 56

BASELINE CHARACTERISTICS:
Arm/Group | Raindrop
Number analyzed (Participants) | 373
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204
  Male | 169
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 290
  African American | 10
  Asian | 6
  Hispanic | 52
  Other | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 373

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Uncorrected Near Visual Acuity (20/40 or Better) in the Implanted Eye
Description: 75% of participants should achieve uncorrected near visual acuity in the implanted eye of 20/40 or better as compared to preoperative baseline
Time Frame: 24 Months
Measure: Number; unit: Count of Participants
Arm/Group | Raindrop
Number analyzed (Participants) | 344
Count of Participants | 336

2. Secondary Outcome: Number of Participants With no or Minimal Loss of Best Corrected Visual Acuity in the Implanted Eye
Description: Less than 5% of participants should lose more than two lines of best corrected distance and near visual acuity in the implanted eye; and less than 1% of participants with preoperative best spectacle corrected visual acuity (BCDVA) of 20/20 in the implanted eye should have best corrected distance and near visual acuity worse than 20/40 in the implanted eye at 6 months postoperative and all subsequent visits.
Time Frame: at 6 months postoperative and all subsequent visits
Population: Numbers analyzed at each timepoint differ due to participant availability
Measure: Number; unit: Count of Participants
Arm/Group | Raindrop
Number analyzed (Participants) | 373
Count of Participants
  # of participants@6M w/loss >/= 2 lines of BCVA: number analyzed (Participants) | 365
  # of participants@6M w/loss >/= 2 lines of BCVA | 0
  # of participants@9M w/loss >/= 2 lines of BCVA: number analyzed (Participants) | 364
  # of participants@9M w/loss >/= 2 lines of BCVA | 1
  # of participants@12M w/loss >/= 2 lines of BCVA: number analyzed (Participants) | 361
  # of participants@12M w/loss >/= 2 lines of BCVA | 1
  # of participants@18M w/loss>/= 2 lines of BCVA: number analyzed (Participants) | 351
  # of participants@18M w/loss>/= 2 lines of BCVA | 1
  # of participant@24M w/loss >/= 2 lines of BCVA: number analyzed (Participants) | 344
  # of participant@24M w/loss >/= 2 lines of BCVA | 1
  # of participants@6M w/BCDVA or BCNVA < 20/40: number analyzed (Participants) | 365
  # of participants@6M w/BCDVA or BCNVA < 20/40 | 0
  # of participants@9M w/BCDVA or BCNVA < 20/40: number analyzed (Participants) | 364
  # of participants@9M w/BCDVA or BCNVA < 20/40 | 1
  # of participants@12M w/BCDVA or BCNVA < 20/40: number analyzed (Participants) | 361
  # of participants@12M w/BCDVA or BCNVA < 20/40 | 0
  # of participants@18M w/BCDVA or BCNVA < 20/40: number analyzed (Participants) | 351
  # of participants@18M w/BCDVA or BCNVA < 20/40 | 0
  # of participants@24M w/BCDVA or BCNVA < 20/40: number analyzed (Participants) | 344
  # of participants@24M w/BCDVA or BCNVA < 20/40 | 0

3. Secondary Outcome: Number of Participants With Induced Manifest Refractive Astigmatism in the Implanted Eye
Description: Less than 5% of participants should have postoperative manifest refractive astigmatism in the implanted eye that increases from baseline by greater than 2.00 D at 6 months postoperative and all subsequent visits.
Time Frame: At 6 months postoperative and all subsequent visits
Population: Numbers analyzed at each timepoint differ due to participant availability.
Measure: Number; unit: Count of Participants
Arm/Group | Raindrop
Number analyzed (Participants) | 373
Count of Participants
  #of participants@6M w/>2D increase in astigmatism: number analyzed (Participants) | 365
  #of participants@6M w/>2D increase in astigmatism | 0
  #of participants@9M w/>2D increase in astigmatism: number analyzed (Participants) | 364
  #of participants@9M w/>2D increase in astigmatism | 0
  #of participants@12M w/>2D increase in astigmatism: number analyzed (Participants) | 361
  #of participants@12M w/>2D increase in astigmatism | 0
  #of participants@18M w/>2D increase in astigmatism: number analyzed (Participants) | 351
  #of participants@18M w/>2D increase in astigmatism | 0
  #of participants@24M w/>2D increase in astigmatism: number analyzed (Participants) | 344
  #of participants@24M w/>2D increase in astigmatism | 0

ADVERSE EVENTS:
Time Frame: Day 1, Week 1, Months 1, 2, 3, 6, 9, 12, 18, 24, 30, 36
Arm/Group | Raindrop
All-Cause Mortality (participants affected / at risk) | 1/373
Serious Adverse Events (participants affected / at risk) | 25/373
Other Adverse Events (participants affected / at risk) | 115/373
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raindrop (N=373)
Death (General disorders) | 1 (1) — Not related to device
Hospitalization due to Ischemic Colitis (Gastrointestinal disorders) | 1 (1) — Non-ocular and not related to device
Hospitalization due to Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Non-ocular and not related to device
Hospitalization due to adverse reaction to medication (General disorders) | 2 (2) — Infection to medication given to treat infection following surgery Seizure, reaction to systemic medication Non-ocular and not related to device
Hospitalization for Transient Ischemic Attack (Nervous system disorders) | 1 (1) — Non-ocular and not related to device
Hospitalization for elevated blood sugar (Blood and lymphatic system disorders) | 1 (1) — Non-ocular and not related to device
Hospitalization for fainting/upper extremity pain - no formal diagnosis (General disorders) | 1 (1) — Non-ocular and not related to device
Hospitalization secondary to heart disease (Cardiac disorders) | 10 (10) — Non-ocular and not related to device
Hospitalization secondary to other surgery (Surgical and medical procedures) | 8 (8) — Transforminal lumbar fusion Cervical fusions with implanted plate and rods Pancreatectomy, Splenectomy (cancer) Gall Bladder removal Nephrectomy Emergency Appendectomy (2) Radical prostatectomy Non-ocular and not related to device
Infection secondary to achilles tendon surgery (Musculoskeletal and connective tissue disorders) | 1 (1) — Non-ocular and not related to device
Melting of the flap (Eye disorders) | 1 (1)
Surgery to repair orbital bone fracture (Eye disorders) | 1 (1) — Relationship to device unknown
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raindrop (N=373)
Ocular infection (Eye disorders) | 7 (8)
Epithelial ingrowth (Eye disorders) | 11 (13)
Loss in BCDVA of > 2 lines (11 letters or more) at 3 months or later (Eye disorders) | 14 (17) — BCDVA = Best Corrected Distance Visual Acuity
Late onset of haze beyond 6 months with loss of 2 lines (10 letters) or more BCVA (Eye disorders) | 4 (4) — BCVA = Best Corrected Visual Acuity
Cataract (with loss in BCDVA greater than or equal to 2 lines at any time (Eye disorders) | 2 (2) — BCDVA = Best Corrected Distance Visual Acuity
Increase in Intraocular Pressure of greater than 10mmHg above baseline (Eye disorders) | 7 (10)
Diffuse Lamellar Keratitis (DLK) (Eye disorders) | 6 (6)
Secondary Surgical Intervention (Eye disorders) | 54 (62) — Inlay Exchange = 18 Inlay Explant = 38 Flap Lift = 4 Cataract Surgery = 1
Posterior Vitreous Detachment (Eye disorders) | 1 (1)
Transient Visual Disturbance (Eye disorders) | 1 (1)
Anterior Uveitis (Eye disorders) | 4 (5)
Corneal Epithelial Defect Involving the Keratectomy (Eye disorders) | 2 (2)
Broken Orbital Bone (Eye disorders) | 1 (1)
Lost, Misaligned, or Misplaced Flap (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agreed to hold this information in confidence and not to disclose it to any third parties for a period of three years from the date of this agreement, or until this information becomes a matter of public knowledge or until a formal agreement for that purpose has been entered into by the parties.